CLINICAL TRIAL: NCT04481737
Title: Peer-delivered and Technology-Assisted Integrated Illness Management and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Harvard University (Other); Vinfen (Industry)
Responsible Party: Principal Investigator, Karen L. Fortuna, Assistant Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D20155
Record Dates: First submitted 2020-07-10; First posted 2020-07-22 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Schizophrenia; Bipolar Disorder; Major Depressive Disorder, Recurrent; Obesity; Cardiovascular Diseases; Diabetes; Smoking; Blood Pressure Disorders; Cholesterol, Elevated
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depressive Disorder, Major; Recurrence; Obesity; Cardiovascular Diseases; Diabetes Mellitus; Smoking; Hypercholesterolemia | interventions — Salvage Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDTA-IIMR (Experimental)
  Interventions: Behavioral: Peer-delivered and Technology Support Integrated Illness Management and Recovery
- Peer support (Active Comparator)
  Interventions: Behavioral: Peer support

INTERVENTIONS:
Behavioral: Peer-delivered and Technology Support Integrated Illness Management and Recovery — PDTA-IIMR is delivered by a peer support specialist with the use of guided IIMR eModules and a smartphone application designed to complement in-person eModule sessions. The eModules are designed to be reviewed with a peer support specialist and consumer during one-hour, weekly, telephonic sessions in a community setting. Each eModule includes videos and experiential learning tasks on psychoeducation and coping skills training.
  Arms: PDTA-IIMR
Behavioral: Peer support — Peer support is a non-manualized form of social support, frequently coupled with instrumental support, that is mutually offered or provided by persons having a mental health condition to others sharing a similar mental health condition to bring about a desired social or personal change. Peer support specialists are provided with 1-hour of supervision each week
  Arms: Peer support

SUMMARY:
Adults with serious mental illness (SMI) are disproportionately affected by medical comorbidity, earlier onset of disease, and 10 to 25 years reduced life expectancy compared to the general population. These high rates of morbidity and early mortality are associated with inadequately managed medical and psychiatric illnesses. A recent systematic review found nine effective self-management interventions that address medical and psychiatric illnesses in adults with SMI. However, there has been limited adoption of these interventions due to both provider and consumer-based factors. Provider-based barriers consist of the lack of an adequate workforce with the capacity, time, and knowledge of effective approaches to self-management support for adults with SMI and chronic health conditions. Consumer-based barriers associated with limited participation in self-management programs include lack of access, engagement, and ongoing community-based support for persons with SMI. Peer support specialists have the potential to address these barriers as they comprise one of the fastest growing sectors of the mental health workforce, have "lived experience" in self-management practices, and offer access to support in the community. However, challenges need to be resolved for peers to be effective providers of evidence-based interventions. For example, peers are frequently trained to provide "peer support" described as "giving and receiving help founded on key principles of respect, shared responsibility, and mutual agreement of what is helpful". Peer support has been associated with increased sense of control, ability to make changes, and decreased psychiatric symptoms. Despite benefits, peer support does not adhere to evidence-based practices for psychiatric and medical self-management and does not follow protocols that ensure fidelity and systematically monitor outcomes. The investigators hypothesize that mobile technology has the potential to overcome these limitations of peer support by providing real-time guidance in fidelity adherent delivery of a peer-delivered, technology-assisted evidence-based self-management intervention (PDTA-IIMR). The investigator will build the necessary expertise to pursue a career developing and testing novel approaches to peer-delivered evidence-based self-management interventions. Training will include: development of peer-delivered interventions; development and design of mobile health-supported interventions; and intervention clinical trials research. Concurrently, this study includes refinement of the intervention protocol with input from peers and consumers and conducting a pilot study evaluating the feasibility and potential effectiveness of PDTA-IIMR compared to routine peer support for N=6 peers and N=40 adults with SMI and chronic health conditions. Outcomes include feasibility, medical and psychiatric self-management skills, functional ability, and mortality risk factors and examine self-efficacy and social support as mechanisms on outcomes.

ELIGIBILITY:
Consumer Inclusion Criteria

Consumer eligibility includes the following:

* (1) participants will be adults age 18 or older who have a chart DSM-V Axis I diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, persistent major depressive disorder (diagnosis will be verified using the Mini-International Neuropsychiatric Interview);
* (2) have been enrolled in treatment for at least 3 months;
* (3) a chart diagnosis of a medical diagnosis of cardiovascular disease, obesity, diabetes, or chronic obstructive pulmonary disease;
* (4) speak and read English; and
* (5) voluntary informed consent for participation in the study by the participant.

Consumer Exclusion Criteria

Consumer participants will be excluded based on the following criteria:

* (1) chart diagnosis of dementia or documented cognitive impairment as indicated by the Mini Mental State Examination score <24;
* (2) major visual, hearing, or motor impairment (measured by potential participants' ability to use a smartphone);
* (3) currently residing in a nursing home;
* (4) terminal illness expected to result of death of participant within one year; or
* (5) consumers with two or more emergency room or hospitalizations in the last 6 months or as determined by the clinical team to be psychiatrically or medically unstable;

Peer Inclusion Criteria

Peer eligibility includes the following:

* (1) Massachusetts certified peer specialist (i.e., to qualify to be a Massachusetts certified peer specialist a person must self-report any mental health diagnosis, be in active treatment, and complete an 80 hour training that includes classes, small group activities, and homework on fundamentals of peer support, cross-cultural partnering, and human experience language. All certified peer specialists must pass a written examination);
* (2) a clinical history of improved psychiatric and medical self-management in the past 6 months;
* (3) speak and read English;
* (4) willing to use technology to deliver an intervention;
* (5) must provide voluntary informed consent for participation in the study; and
* (6) have worked as a certified peer specialist with people with SMI for 1+ years.

Peer Exclusion Criteria

Peer participants will be excluded based on the following criteria:

* (1) chart diagnosis of dementia or documented cognitive impairment as indicated by the Mini Mental State Examination score <24;
* (2) major visual, hearing, or motor impairment (measured by potential participants' ability to use a tablet); and
* (3) certified peer specialists with two or more emergency room or hospitalizations in the last 6 months or as determined by the clinical team to be psychiatrically or medically unstable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Change in number of study drop-outs, attendance, and adherence from baseline to 3-months | Baseline and 3-months
  Review case notes written by peer support specialists to examine count data on attrition, attendance, and patient adherence.
Change in average fidelity scores | Baseline and 3-months
  Peer Support specialists will independently rate themselves after each session using the PDTA-IIMR fidelity scale. The standards used for establishing the items and ratings were determined by expert sources and empirical research.

SECONDARY OUTCOMES:
Change from baseline mortality risk index to 3-months and 6-month follow-up | Baseline, 3-months, and 6-months
  Avoidable Mortality Risk Index includes an examination of modifiable risk factors include: smoking; high blood pressure; excess body weight; high blood glucose; high cholesterol; high alcohol intake; low physical activity; poor diet.
Change from baseline self efficacy to 3-months and 6-month follow-up | Baseline, 3-months, and 6-months
  Self-Efficacy for Managing Chronic Disease. Self-Efficacy for Managing Chronic Disease is a six-item scale that assesses domains of self-efficacy: symptom control, role function, emotional functioning, and communicating with physicians. Higher scores indicate greater self-efficacy.
Change from baseline social support to 3-months and 6-month follow-up | Baseline, 3-months, and 6-months
  Medical Outcomes Study Social Support Survey. Medical Outcomes Study Social Support is a 19-item scale that assesses domains of social support: emotional/informational, tangible, affection, and positive social interaction. Higher scores indicate higher levels of social support.
Change from baseline mental health self-management skills to 3-months and 6-month follow-up | Baseline, 3-months, and 6-months
  Illness Management and Recovery Scale. The Illness Management and Recovery Scale is a valid, reliable 15-item scale that assesses domains of illness management. Each item addresses psychiatric illness, management, and recovery. Higher scores equate to higher ability to manage psychiatric conditions.
Change from baseline medical self-management skills to 3-months and 6-month follow-up | Baseline, 3-months, and 6-months
  Self-Rated Abilities for Health Practices Scale.The Self-Rated Abilities for Health Practices Scale is a 28-item scale that assesses confidence to execute health practices that has shown reliability and validity with adults with disabilities. This scale includes four subscales: exercise, nutrition, responsible health practice, and psychological well-being. Higher scores indicate higher levels of self-efficacy.
Change from baseline functional ability to 3-months and 6-month follow-up | Baseline, 3-months, and 6-months
  PROMIS Global Health. The PROMIS Global Health includes 10-items that measures five core PROMIS domains (physical function, pain, fatigue, emotional distress, social health). The measure is agnostic, rather than disease-specific, and commonly used to show an individuals' assessment of their overall health. Higher scores indicate better functional ability.
Change from baseline disability to 3-months and 6-month follow-up | Baseline, 3-months, and 6-months
  London Handicap Scale. The London Handicap Scale measures health status and includes domains of independent living skills: mobility, physical independence, occupation, social integration, orientation, and economic self-sufficiency. Higher scores indicate better functional ability.
Change from baseline level of cardiovascular disease risk to 3-months and 6-month follow-up | Baseline, 3-months, and 6-months
  Framingham Risk Score. Framingham Risk Score includes risk factors: age; sex; LDL cholesterol; HDL cholesterol; blood pressure; diabetes; and smoking. A higher score indicates worse outcomes.

OTHER OUTCOMES:
Change from baseline level of loneliness to 3-months and 6-month follow-up | Baseline, 3-months, and 6-months
  UCLA Loneliness Scale. For loneliness each of the three-item version of the UCLA Loneliness Scale are rated on a four-point scale, with higher values indicative of greater loneliness. Items asked about how often individuals felt left out and isolated from others, and how often they felt that there are people that really understand them or that they can talk to.
Change from baseline patient satisfaction to 3-months and 6-month follow-up | Baseline, 3-months, and 6-months
  Adult Patient Satisfaction Survey. The 36-item Adult Patient Satisfaction Survey designed to measure patient satisfaction in receiving mental health services in a community-based mental health system. Higher scores indicate greater patient satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Vinfen, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Tools (data, assays, libraries, research tools, reagents, model organisms, etc.) will be made available, in accordance with the NIH Data Sharing Policy (http://grants.nih.gov/grants/policy/data_sharing) and Model Organism Sharing Policy (http://grants.nih.gov/grants/policy/model_organism/index.htm), to all researchers in both the private and public sector free or for a nominal charge and with minimal restriction. In some cases the Trustees of Dartmouth College (the institution) may determine that the public and the research community are better served by a licensing program whether or not patents have been filed. This may be relevant, for example, if a tool is best distributed under license to guarantee reagent availability and quality.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Fortuna KL, Cui S, Lebby S, Xie H, Bruce ML, Bartels SJ. PeerTECH: a randomized controlled trial of a peer-led mobile health intervention to improve medical and psychiatric self-management for persons with serious mental illness. Mhealth. 2025 Jun 30;11:28. doi: 10.21037/mhealth-24-64. eCollection 2025. PMID 40755935